CLINICAL TRIAL: NCT07014332
Title: Comparison of Alignment Efficiency of Steel Vs Elastomeric Ligatures In Lower Anterior Teeth: A Randomized Clinical Trial
Brief Title: Comparison of Alignment Efficiency of Steel Vs Elastomeric Ligatures In Lower Anterior Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber College of dentistry (Other)
Responsible Party: Principal Investigator, Aatikah Javaid, Principal investigator, Khyber College of dentistry
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 45/ADR/KCD
Record Dates: First submitted 2025-05-21; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Malocclusion of Anterior Teeth
Keywords: Orthodontic treatment; Ligature type; Steel ligature; Elastomeric ligature; Alignment time

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Group A received steel ligature and group B elastomeric ligature (Other)
  Interventions: Device: Steel ligature; Device: Elastomeric ligature

INTERVENTIONS:
Device: Steel ligature — Steel ligatures that are used to ligate wire with bracket
Device: Elastomeric ligature — Elastomeric ligature that is used to ligate wire to bracket

SUMMARY:
To compare the treatment time required by elastomeric ligatures and steel ligatures, in days, to achieve complete alignment of the lower anterior teeth.

DETAILED DESCRIPTION:
Treatment time required to achieve alignment by two ligation methods will help us in future to choose a better method. The two methods study are elastomeric ligature and steel ligature.

ELIGIBILITY:
Inclusion Criteria:

1. Patients coming for fixed orthodontic treatment requiring premolar extraction in mandibular arch.
2. Age 12-18 years.
3. No adjunct therapeutic intervention involving functional or orthopaedic appliances.
4. Little's Irregularity index score of 7-9mm.

Exclusion Criteria:

1. Patients with systemic conditions and taking medications affecting tooth movement.
2. Lower anterior teeth that are missing, impacted or unerupted, or have fractured crown, restorations, Enamel Defects, Caries.
3. Poor periodontal health

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Actual)
Dates: Start 2024-09-19 (Actual); Primary Completion 2025-05-10 (Actual); Study Completion 2025-05-10 (Actual)

PRIMARY OUTCOMES:
Alignment time to reach little irregularity index of zero | From recruitment to 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Ahsan Mehmood Shah, Fellowship, Study Director — Khyber College of dentistry
Locations (1):
- Khyber College of Dentistry, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-09): https://cdn.clinicaltrials.gov/large-docs/32/NCT07014332/Prot_SAP_000.pdf
  • Informed Consent Form (2024-09-19): https://cdn.clinicaltrials.gov/large-docs/32/NCT07014332/ICF_001.pdf